CLINICAL TRIAL: NCT06248671
Title: EpisodicStatinMig. A Multicentre, Triple Blind, Placebo Controlled, Parallel Group Study of Atorvastatin in Episodic Migraine
Brief Title: Prophylactic Treatment With Atorvastatin for Episodic Migraine.
Acronym: EStatinMig
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Haukeland University Hospital (Other); Oslo University Hospital (Other); University Hospital of North Norway (Other); University Hospital, Akershus (Other); Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-502176-23-01
Record Dates: First submitted 2024-01-19; First posted 2024-02-08 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Episodic Migraine
Keywords: Migraine; Atorvastatin; Randomized controlled trial
MeSH Terms: conditions — Migraine Disorders | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Parallel group study with three arms, comparing Atorvastatin 20 mg and 40 mg against placebo. Each participant will receive 84 encapsulated tablets. The participant will take one capsule orally each day, preferably at the same time of the day.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blind (blinded to patients, study personnel, and statistician).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Atorvastatin 40mg (Active Comparator): Each participant in this arm will receive 40mg atorvastatin once daily for 84 days.
  Interventions: Drug: Atorvastatin 40mg
- Atorvastatin 20mg (Active Comparator): Each participant in this arm will receive 20mg atorvastatin once daily for 84 days.
  Interventions: Drug: Atorvastatin 20mg
- Placebo (Placebo Comparator): Each participant in this arm will receive placebo once daily for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 40mg — Each tablet will be taken once daily for 84 days.
  Other Names: Lipitor
  Arms: Atorvastatin 40mg
Drug: Placebo — Each tablet will be taken once daily for 84 days
  Arms: Placebo
Drug: Atorvastatin 20mg — Each tablet will be taken once daily for 84 days.
  Other Names: Lipitor
  Arms: Atorvastatin 20mg

SUMMARY:
The main objective of this study is to see whether the favorable preventative effect of Atorvastatin 40mg per day in episodic migraine, that was found previously in three smaller randomized controlled cross-over studies, can be confirmed in a larger, multicenter, randomized controlled parallel group study. In addition it will be investigated whether 1) there is an effect of a daily dose of 20mg Atorvastatin, 2) whether the favorable side effect profile, seen in previous studies, can be confirmed, and whether it is even better with the smaller dose, and 3) estimating the cost of Atorvastatin treatment, considering cost of medicine, cost of acute attack medicine, and cost of lost worktime.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* Signed informed consent.
* Episodic migraine with or without aura according to ICHD-3 criteria.
* At inclusion, patients should retrospectively have from 4 to 14 migraine attacks per month during the last 3 months. This frequency must be confirmed in the headache diary before randomisation to treatment.
* Debut of migraine at least one year prior to inclusion based on information in the patient record or by careful examination of previous headache history.
* Start of migraine before 50 years.
* No use of other migraine prophylactics during the study.
* For women of child-bearing potential, there must be no pregnancy or planned pregnancy during the study period, and use of highly effective contraception.

After the baseline period, just before randomisation to the study drug, inclusion criteria will be evaluated once more, and the headache diary will be evaluated. If there are, according to the headache diary, fewer attacks than 4 or more than 14 per month, the baseline period can be extended to 8 weeks, and the patient can be randomized to a treatment then if there is a mean of 4-14 attacks per 4 weeks during the 8-week's period.

Exclusion Criteria:

* Interval headache not distinguishable from migraine.
* Chronic migraine, chronic tension-type headache, medication overuse headache or other headache occurring on ≥ 15 days/month.
* Pregnancy, planning to get pregnant, inability to use contraceptives, and lactating.
* Clinical information on or signs of cholestasis or decreased hepatic or renal function.
* High degree of comorbidity and/or frailty associated with reduced life expectancy or high likelihood of hospitalization, at the discretion of the investigator.
* Hypersensitivity to statins or previous use of statins.
* History of angioneurotic oedema.
* Use of medicines for migraine prophylaxis less than 4 weeks, or of botulinum toxin less than 16 weeks, prior to start of study.
* Current use of antiviral treatment against hepatitis C.
* Significant psychiatric illness.
* Having tried ≥ 3 prophylactic drugs against migraine during the last 10 years.
* Requiring detoxification from acute medication (triptans, opioids).
* Consistently failing to respond to any acute migraine medication.
* Alcohol or illicit drug dependence.
* Inability to understand study procedures and to comply with them for the entire length of the study.
* Treatment for hypothyroidism.
* Lactose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of migraine days | 4 weeks
  Change in number of migraine days/4 weeks from the baseline period to the treatment period.

SECONDARY OUTCOMES:
Number of responders | 12 weeks
  Number of responders (≥ 50% improvement from baseline)
Rate of adverse events | 12 weeks
  Number of patients with adverse events
Number of doses with acute medication | 12 weeks
  Doses of triptans or analgesics per 4 weeks
Number of days with sick leave | 12 weeks
  Days with sick leave per 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marte-Helene Bjørk, Professor, Principal Investigator — Haukeland University Hospital; Kjersti G Vetvik, Ph.d., Principal Investigator — University Hospital, Akershus; Bendik S Winsvold, Post.doc., Principal Investigator — Oslo University Hospital, Ullevål; Anne H Aamodt, Senior researcher, Principal Investigator — Oslo University Hospital; Lise R Øie, Post.doc., Principal Investigator — St. Olavs Hospital; Linn H Steffensen, Associate Professor II, Principal Investigator — University Hospital Northern Norway
Locations (6):
- Norway (6):
  - Haukeland University Hospital, Bergen
  - University Hospital, Akershus, Lørenskog
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Oslo University Hospital, Ullevål, Oslo
  - University Hospital Northern Norway, Tromsø
  - St. Olavs hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steiner TJ, Stovner LJ, Jensen R, Uluduz D, Katsarava Z; Lifting The Burden: the Global Campaign against Headache. Migraine remains second among the world's causes of disability, and first among young women: findings from GBD2019. J Headache Pain. 2020 Dec 2;21(1):137. doi: 10.1186/s10194-020-01208-0. No abstract available. PMID 33267788
- [Background] Stovner LJ, Hagen K, Linde M, Steiner TJ. The global prevalence of headache: an update, with analysis of the influences of methodological factors on prevalence estimates. J Headache Pain. 2022 Apr 12;23(1):34. doi: 10.1186/s10194-022-01402-2. PMID 35410119
- [Background] Evers S, Afra J, Frese A, Goadsby PJ, Linde M, May A, Sandor PS; European Federation of Neurological Societies. EFNS guideline on the drug treatment of migraine--revised report of an EFNS task force. Eur J Neurol. 2009 Sep;16(9):968-81. doi: 10.1111/j.1468-1331.2009.02748.x. PMID 19708964
- [Background] Langohr HD, Gerber WD, Koletzki E, Mayer K, Schroth G. Clomipramine and metoprolol in migraine prophylaxis--a double-blind crossover study. Headache. 1985 Mar;25(2):107-13. doi: 10.1111/j.1526-4610.1985.hed2502107.x. No abstract available. PMID 3886599
- [Background] Ziegler DK, Hurwitz A, Hassanein RS, Kodanaz HA, Preskorn SH, Mason J. Migraine prophylaxis. A comparison of propranolol and amitriptyline. Arch Neurol. 1987 May;44(5):486-9. doi: 10.1001/archneur.1987.00520170016015. PMID 3579659
- [Background] Tronvik E, Stovner LJ, Helde G, Sand T, Bovim G. Prophylactic treatment of migraine with an angiotensin II receptor blocker: a randomized controlled trial. JAMA. 2003 Jan 1;289(1):65-9. doi: 10.1001/jama.289.1.65. PMID 12503978
- [Background] Stovner LJ, Linde M, Gravdahl GB, Tronvik E, Aamodt AH, Sand T, Hagen K. A comparative study of candesartan versus propranolol for migraine prophylaxis: A randomised, triple-blind, placebo-controlled, double cross-over study. Cephalalgia. 2014 Jun;34(7):523-32. doi: 10.1177/0333102413515348. Epub 2013 Dec 11. PMID 24335848
- [Background] Mei D, Capuano A, Vollono C, Evangelista M, Ferraro D, Tonali P, Di Trapani G. Topiramate in migraine prophylaxis: a randomised double-blind versus placebo study. Neurol Sci. 2004 Dec;25(5):245-50. doi: 10.1007/s10072-004-0350-0. PMID 15624081
- [Background] Brandes JL, Saper JR, Diamond M, Couch JR, Lewis DW, Schmitt J, Neto W, Schwabe S, Jacobs D; MIGR-002 Study Group. Topiramate for migraine prevention: a randomized controlled trial. JAMA. 2004 Feb 25;291(8):965-73. doi: 10.1001/jama.291.8.965. PMID 14982912
- [Background] Bulut S, Berilgen MS, Baran A, Tekatas A, Atmaca M, Mungen B. Venlafaxine versus amitriptyline in the prophylactic treatment of migraine: randomized, double-blind, crossover study. Clin Neurol Neurosurg. 2004 Dec;107(1):44-8. doi: 10.1016/j.clineuro.2004.03.004. PMID 15567552
- [Background] Couch JR; Amitriptyline Versus Placebo Study Group. Amitriptyline in the prophylactic treatment of migraine and chronic daily headache. Headache. 2011 Jan;51(1):33-51. doi: 10.1111/j.1526-4610.2010.01800.x. Epub 2010 Nov 10. PMID 21070231
- [Background] Sacco S, Bendtsen L, Ashina M, Reuter U, Terwindt G, Mitsikostas DD, Martelletti P. Correction to: European headache federation guideline on the use of monoclonal antibodies acting on the calcitonin gene related peptide or its receptor for migraine prevention. J Headache Pain. 2019 May 23;20(1):58. doi: 10.1186/s10194-019-0972-5. PMID 31122188
- [Background] Katsarava Z, Mania M, Lampl C, Herberhold J, Steiner TJ. Poor medical care for people with migraine in Europe - evidence from the Eurolight study. J Headache Pain. 2018 Feb 1;19(1):10. doi: 10.1186/s10194-018-0839-1. PMID 29392600
- [Background] Buettner C, Nir RR, Bertisch SM, Bernstein C, Schain A, Mittleman MA, Burstein R. Simvastatin and vitamin D for migraine prevention: A randomized, controlled trial. Ann Neurol. 2015 Dec;78(6):970-81. doi: 10.1002/ana.24534. Epub 2015 Nov 13. PMID 26418341
- [Background] Hesami O, Sistanizad M, Asadollahzade E, Johari MS, Beladi-Moghadam N, Mazhabdar-Ghashghai H. Comparing the Effects of Atorvastatin With Sodium Valproate (Divalproex) on Frequency and Intensity of Frequent Migraine Headaches: A Double-blind Randomized Controlled Study. Clin Neuropharmacol. 2018 May/Jun;41(3):94-97. doi: 10.1097/WNF.0000000000000280. PMID 29746282
- [Background] Ganji R, Majdinasab N, Hesam S, Rostami N, Sayyah M, Sahebnasagh A. Does atorvastatin have augmentative effects with sodium valproate in prevention of migraine with aura attacks? A triple-blind controlled clinical trial. J Pharm Health Care Sci. 2021 Apr 1;7(1):12. doi: 10.1186/s40780-021-00198-8. PMID 33789774
- [Background] Sherafat A, Sahebnasagh A, Rahmany R, Mohammadi F, Saghafi F. The preventive effect of the combination of atorvastatin and nortriptyline in migraine-type headache: a randomized, triple-blind, placebo-controlled trial. Neurol Res. 2022 Apr;44(4):311-317. doi: 10.1080/01616412.2021.1981105. Epub 2022 Jan 17. PMID 35037597
- [Background] Endo A. The discovery and development of HMG-CoA reductase inhibitors. J Lipid Res. 1992 Nov;33(11):1569-82. No abstract available. PMID 1464741
- [Background] Musial J, Undas A, Gajewski P, Jankowski M, Sydor W, Szczeklik A. Anti-inflammatory effects of simvastatin in subjects with hypercholesterolemia. Int J Cardiol. 2001 Feb;77(2-3):247-53. doi: 10.1016/s0167-5273(00)00439-3. PMID 11182189
- [Background] Yanuck D, Mihos CG, Santana O. Mechanisms and clinical evidence of the pleiotropic effects of the hydroxy-methyl-glutaryl-CoA reductase inhibitors in central nervous system disorders: a comprehensive review. Int J Neurosci. 2012 Nov;122(11):619-29. doi: 10.3109/00207454.2012.704455. Epub 2012 Aug 14. PMID 22720798
- [Background] Zhou Q, Liao JK. Pleiotropic effects of statins. - Basic research and clinical perspectives -. Circ J. 2010 May;74(5):818-26. doi: 10.1253/circj.cj-10-0110. Epub 2010 Apr 15. PMID 20424337
- [Background] Salagre E, Fernandes BS, Dodd S, Brownstein DJ, Berk M. Statins for the treatment of depression: A meta-analysis of randomized, double-blind, placebo-controlled trials. J Affect Disord. 2016 Aug;200:235-42. doi: 10.1016/j.jad.2016.04.047. Epub 2016 Apr 27. PMID 27148902
- [Background] Millar PJ, Floras JS. Statins and the autonomic nervous system. Clin Sci (Lond). 2014 Mar;126(6):401-15. doi: 10.1042/CS20130332. PMID 24274967
- [Background] Lennernas H. Clinical pharmacokinetics of atorvastatin. Clin Pharmacokinet. 2003;42(13):1141-60. doi: 10.2165/00003088-200342130-00005. PMID 14531725
- [Background] Jones PH, Davidson MH, Stein EA, Bays HE, McKenney JM, Miller E, Cain VA, Blasetto JW; STELLAR Study Group. Comparison of the efficacy and safety of rosuvastatin versus atorvastatin, simvastatin, and pravastatin across doses (STELLAR* Trial). Am J Cardiol. 2003 Jul 15;92(2):152-60. doi: 10.1016/s0002-9149(03)00530-7. PMID 12860216
- [Background] Diener HC, Tassorelli C, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ, Houle TT, Hoek TCVD, Martinelli D, Terwindt GM; International Headache Society Clinical Trials Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of migraine attacks in episodic migraine in adults. Cephalalgia. 2020 Sep;40(10):1026-1044. doi: 10.1177/0333102420941839. Epub 2020 Jul 28. PMID 32722936
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Buettner C, Burstein R. Association of statin use and risk for severe headache or migraine by serum vitamin D status: a cross-sectional population-based study. Cephalalgia. 2015 Aug;35(9):757-66. doi: 10.1177/0333102414559733. Epub 2014 Nov 25. PMID 25424706
- [Background] Finegold JA, Manisty CH, Goldacre B, Barron AJ, Francis DP. What proportion of symptomatic side effects in patients taking statins are genuinely caused by the drug? Systematic review of randomized placebo-controlled trials to aid individual patient choice. Eur J Prev Cardiol. 2014 Apr;21(4):464-74. doi: 10.1177/2047487314525531. Epub 2014 Mar 12. PMID 24623264
- [Background] Gupta A, Thompson D, Whitehouse A, Collier T, Dahlof B, Poulter N, Collins R, Sever P; ASCOT Investigators. Adverse events associated with unblinded, but not with blinded, statin therapy in the Anglo-Scandinavian Cardiac Outcomes Trial-Lipid-Lowering Arm (ASCOT-LLA): a randomised double-blind placebo-controlled trial and its non-randomised non-blind extension phase. Lancet. 2017 Jun 24;389(10088):2473-2481. doi: 10.1016/S0140-6736(17)31075-9. Epub 2017 May 2. PMID 28476288
- [Background] Jenssen AB, Stovner LJ, Tronvik E, Sand T, Helde G, Gravdahl GB, Hagen K. The crossover design for migraine preventives: an analyses of four randomized placebo-controlled trials. J Headache Pain. 2019 Dec 27;20(1):119. doi: 10.1186/s10194-019-1067-z. PMID 31881823
- See also: Statins rarely cause adverse effects — https://tidsskriftet.no/2022/01/kronikk/statiner-gir-sjelden-bivirkninger
- See also: Treatment with statins — https://tidsskriftet.no/2013/06/legemidler-i-praksis/behandling-med-statiner
- See also: Serendipity atorvastatin and vitamin D — https://www.australianpharmacist.com.au/old-drug-new-indication-statins-and-vitamin-d-for-migraines/

DOCUMENTS (2):
  • Study Protocol (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT06248671/Prot_004.pdf
  • Informed Consent Form (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT06248671/ICF_005.pdf